CLINICAL TRIAL: NCT06553508
Title: Trochanteric Bursal Repair After a Total Hip Replacement - Are There Benefits During the First 90 Days
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Principal Investigator, Enejd Veizi, MD, Assistant Professor, Ankara City Hospital Bilkent
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: E2-21-1124
Record Dates: First submitted 2024-08-12; First posted 2024-08-14 (Actual); Last update posted 2024-08-16 (Actual); Status verified 2024-08

CONDITIONS: Bursa; Tuberculous; Hip Bursitis; Deep Gluteal Syndrome; Hip Disease
Keywords: bursa; greater trochanter; hip arthroplasty; deep gluteal syndrome; piriformis syndrome
MeSH Terms: conditions — Latent Tuberculosis; Hip socket neuropathy; Piriformis Muscle Syndrome

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Unrepaired bursa group (Active Comparator): As a routine procedure in our centre, the trochanteric bursa is left unrepaired after a hip arthroplasty. The conventional joint closure is performed after reduction and the layers are closed in a routine fashion.
  Interventions: Procedure: Trochanteric bursa unrepaired
- Repaired Bursa group (Experimental): For the experimental arm, the trochanteric bursa is repaired after a hip arthroplasty. The conventional joint closure is performed after reduction and then the bursa is retrieved and repaired. Layers are then closed in a routine fashion.
  Interventions: Procedure: Trochanteric bursa repaired

INTERVENTIONS:
Procedure: Trochanteric bursa repaired — As a routine procedure in our centre, the trochanteric bursa is left unrepaired after a hip arthroplasty.
  Arms: Repaired Bursa group
Procedure: Trochanteric bursa unrepaired — For the experimental arm, the trochanteric bursa is repaired after a hip arthroplasty. The conventional joint closure is performed after reduction and then the bursa is retrieved and repaired.
  Arms: Unrepaired bursa group

SUMMARY:
During total hip arthroplasty surgery, the trochanteric bursa is routinely excised. This anatomical structure, which functions as a soft tissue barrier, is generally recommended for removal as it facilitates the surgical approach. However, recent studies have suggested that the trochanteric bursa is an important soft tissue barrier and may protect against infections. The aim of this study is to evaluate the differences in infection rates, wound complications, deep gluteal syndrome presence, pain, and clinical scores within the first 90 days between patients in whom the trochanteric bursa was repaired and those in whom it was not, and to provide recommendations regarding bursal repair.

DETAILED DESCRIPTION:
During total hip arthroplasty surgery, the trochanteric bursa is routinely excised. This anatomical structure, which functions as a soft tissue barrier, is typically recommended for removal as it facilitates the surgical approach. However, recent studies have suggested that the trochanteric bursa is an important soft tissue barrier and may provide protection against infections. The aim of this study is to evaluate the differences in infection rates, wound complications, deep gluteal syndrome presence, pain, and clinical scores within the first 90 days between patients in whom the trochanteric bursa was repaired and those in whom it was not, and to provide recommendations regarding bursal repair.

This research will be a prospective randomized controlled trial with patients subjected to sequential randomization. One group of patients will undergo the routine excision of the bursa during surgery, referred to as Group 1. In the other group, the trochanteric bursa will be carefully retracted and subsequently repaired in its anatomical location beneath the fascia after the surgical procedure. Wound closure will be performed routinely, with subcutaneous and skin closure. All patients will have a Hemovac drain placed, and they will follow the same rehabilitation protocol.

Patients will be evaluated on postoperative days15, 30, and 90 using Visual Analog Scale scores, and on days 30 and 90 using the Harris Hip Score. Additionally, patients will be assessed for tenderness on palpation, the presence of hip snapping (a sensation of the hip catching), hemoglobin drop, 90-day infection rates, and the presence of deep gluteal syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Patients between 18 to 90 years of age
* With a diagnosis of primary hip osteoarthritis
* Willing to be included in the study

Exclusion Criteria:

* Patients who had a known history of trochanteric bursitis, deep gluteal syndrome, sciatica, vertebral fracture, hip fracture, hip arthroscopy, and core decompression surgery
* Patients who had a history of bursal injection within 6 months
* Patients undergoing hip arthroplasty with a shortening osteotomy

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-01-01 (Actual)

PRIMARY OUTCOMES:
Rate of superficial wound problems | First postoperative 90 days
  Wound leakage, superficial infection, wound dehiscence - Recorded as Yes / No
Rate of posterior gluteal pain | First postoperative 90 days
  The condition is also refered to as Deep Gluteal Syndrome - Recorded as Yes / No
Rate of painful trochanteric bursitis | First postoperative 90 days
  Recorded as pain on the trochanteric region on palpation - Recorded as Yes / No

SECONDARY OUTCOMES:
Range of motion (ROM) | First postoperative 90 days
  Angular measurement of hip joint motion - minimum value:0, maximum value 130, higher values mean better outcome
Visual Analog Scale (VAS) | First postoperative 90 days
  minimum value:0, maximum value 10, higher values mean worse outcome
Harris Hip Score (HHS) | First postoperative 90 days
  minimum value:0, maximum value 100, higher values mean better outcome

CONTACTS AND LOCATIONS:
Overall Officials: Enejd Veizi, MD, Principal Investigator — Ankara City Hospital Bilkent
Locations (1):
- Ankara Bilkent City Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Schwartsmann CR, Loss F, de Freitas Spinelli L, Furian R, Silva MF, Zanatta JM, Boschin LC, Goncalves RZ, Yepez AK. Association between trochanteric bursitis, osteoarthrosis and total hip arthroplasty. Rev Bras Ortop. 2014 Apr 25;49(3):267-70. doi: 10.1016/j.rboe.2014.04.009. eCollection 2014 May-Jun. PMID 26229811
- [Background] Shemesh SS, Moucha CS, Keswani A, Maher NA, Chen D, Bronson MJ. Trochanteric Bursitis Following Primary Total Hip Arthroplasty: Incidence, Predictors, and Treatment. J Arthroplasty. 2018 Apr;33(4):1205-1209. doi: 10.1016/j.arth.2017.11.016. Epub 2017 Nov 13. PMID 29195847
- [Background] Moerenhout K, Benoit B, Gaspard HS, Rouleau DM, Laflamme GY. Greater trochanteric pain after primary total hip replacement, comparing the anterior and posterior approach: A secondary analysis of a randomized trial. Orthop Traumatol Surg Res. 2021 Dec;107(8):102709. doi: 10.1016/j.otsr.2020.08.011. Epub 2020 Oct 31. PMID 33132093